CLINICAL TRIAL: NCT04151290
Title: Cognoa ASD Diagnosis Aid Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cognoa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Q170886
Record Dates: First submitted 2019-10-09; First posted 2019-11-05 (Actual); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: All subjects will undergo both investigational and comparator diagnosis for ASD.
Masking Description: All participants and healthcare providers will be blinded to the diagnosis results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cognoa Assessment (Experimental): Cognoa diagnostic ASD device.
  Interventions: Diagnostic Test: Cognoa ASD diagnostic device

INTERVENTIONS:
Diagnostic Test: Cognoa ASD diagnostic device — Cognoa device is intended to aid healthcare providers in diagnosing Autism Spectrum Disorder (ASD)

SUMMARY:
The primary objective of this study is to collect data to ascertain the Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of the current version of the Cognoa diagnostic device.

DETAILED DESCRIPTION:
To assess the ability of the diagnostic device to aid in the diagnosis of ASD by comparing its diagnostic output with the clinical reference standard, consisting of a diagnosis made by a specialist clinician, based on DSM-5 criteria and validated by one or more reviewing specialist clinicians

ELIGIBILITY:
General Inclusion Criteria:

* Caregiver must be able to read, understand and sign the Informed Consent Form (ICF).
* Caregiver or HCP concern for developmental delay.
* Female or Male, >18 to <72 months of age

General Exclusion Criteria:

* Subjects with a prior diagnosis of ASD rendered by a healthcare professional.
* Subjects whose age on the date of enrollment is outside the target age range.
* Subjects or caregivers who have been previously enrolled in any Cognoa clinical study or survey.

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 711 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharief Taraman, MD, Study Director — Cognoa, Inc.
Locations (16):
- United States (16):
  - Melmed Center, Scottsdale, Arizona
  - The Nicholls Group, Scottsdale, Arizona
  - Orange County Child Neurology, Laguna Niguel, California
  - Pediatric Neurology of Orange County, Laguna Niguel, California
  - Private Practice, Laguna Niguel, California
  - Private Practice, Los Angeles, California
  - Private Practice, Palo Alto, California
  - MediSync Clinical Research Hattiesburg Clinic, Petal, Mississippi
  - PriMed Clinical Research, Dayton, Ohio
  - ARC Clinical Research at Wilson Parke, Austin, Texas
  - ARC Clinical Research William Cannon, Austin, Texas
  - ARC Clinical Research Kelly Lane, Pflugerville, Texas
  - Texas Child Neurology, Plano, Texas
  - Private Practice, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Multicare Health System - Mary Bridge Pediatrics, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognoa Assessment
Started | 711
Completed | 425
Not Completed | 286
Not completed — The COVID-19 Pandemic made it hard for subjects to complete the study. | 286

BASELINE CHARACTERISTICS:
Population: Children ages 18-72 months
Arm/Group | Cognoa Assessment
Number analyzed (Participants) | 425
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 425
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.3 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 271
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race\Ethnicity: American Indian only | 0
  Race\Ethnicity: Asian only | 18
  Race\Ethnicity: Black only | 56
  Race\Ethnicity: Hawaiian or Pacific Islander only | 1
  Race\Ethnicity: Hispanic or Latino or Latino only | 49
  Race\Ethnicity: Multiple races and/or ethnicities indicated | 57
  Race\Ethnicity: Non-Hispanic White only | 229
  Race\Ethnicity: Other race indicated only | 5
  Race\Ethnicity: Unknown | 10

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Predictive Value of ASD Dx in Relation to Clinician Diagnostic Evaluation
Description: Achievement of a composite of positive predictive value (PPV) greater than 65% and negative predictive value (NPV) greater than 85% for the device in relation to the clinical reference standard in the overall study population:
Time Frame: 6 Weeks
Population: Participants
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Cognoa Assessment
Number analyzed (Participants) | 425
percent
  PPV | 80.8 [70.3 to 88.8]
  NPV | 98.3 [90.6 to 100]

2. Primary Outcome: No Result Percentage
Description: Measurement of the percentage of children for whom the device has provided no result.
Time Frame: 6 Weeks
Population: Participants
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Cognoa Assessment
Number analyzed (Participants) | 425
percent | 68.2 [63.6 to 72.6]

3. Secondary Outcome: Device Sensitivity and Specificity
Description: Sensitivity and Specificity of the device in relation to the clinical reference standard in the overall study population.
Time Frame: 6 Weeks
Population: Participants
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Cognoa Assessment
Number analyzed (Participants) | 425
percent
  Sensitivity | 51.6 [42.4 to 60.8]
  Specificity | 18.5 [14.3 to 23.3]

ADVERSE EVENTS:
Time Frame: Just over 1 year.
Description: There were no difference in definitions used to collect adverse event information from those provided from clinicaltrials.gov
Arm/Group | Cognoa Assessment
All-Cause Mortality (participants affected / at risk) | 0/425
Serious Adverse Events (participants affected / at risk) | 0/425
Other Adverse Events (participants affected / at risk) | 0/425

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pub./disc. of the Study(30)days prior to submission for pub./disc. Sponsor to review/comment on the proposed pub./disc. identify any Confidential Information of Sponsor to be deleted from the proposed pub./disc.; protect proprietary rights to Inventions. Sponsor shall provide comments or identify any Confidential Information to be deleted from the proposed pub./disc.(30)day period.Upon Sponsor's reasonable request prior to expiration of the initial thirty (30) day review,Investigator shall delay

DOCUMENTS (2):
  • Study Protocol (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT04151290/Prot_004.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT04151290/SAP_005.pdf